CLINICAL TRIAL: NCT05397652
Title: Effects of the Application of a New Pharmacological Protocol for Shoulder Arthroscopy in Beach Chair Position
Brief Title: The Aim of This Study is to Examine the Effect of Intravenously Administered Tranexamic Acid (TXA) on the Visual Clarity, Perioperative Hemorrhage, Duration and Early Postoperative Course of Shoulder Arthroscopy in Beach Chair Position.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nikola Matejcic (Other)
Collaborators: University orthopaedic and trauma hospital Lovran (Unknown); University of Rijeka, The Faculty of Medicine (Unknown); University of Zagreb, The Faculty of Kinesiology (Unknown)
Responsible Party: Sponsor-Investigator, Nikola Matejcic, Principal investigator, Clinic for Orthopedics Lovran
Organization: Clinic for Orthopedics Lovran (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MATTXA2022
Record Dates: First submitted 2022-05-18; First posted 2022-05-31 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Rotator Cuff Tears; Hemorrhage, Surgical; Shoulder Injuries
Keywords: Arthroscopy; Hemorrhage; Shoulder; Tranexamic acid
MeSH Terms: conditions — Rotator Cuff Injuries; Blood Loss, Surgical; Shoulder Injuries; Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic acid injectable product (Experimental): Patients from the experimental group will receive 10 minutes before the procedure 1 g of tranexamic acid in 100 ml of saline intravenously
  Interventions: Drug: Tranexamic Acid Injectable Product
- Placebo (Placebo Comparator): Patients from the control group will receive 10 minutes before the procedure 100 ml sterile saline intravenously
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid Injectable Product — Patients from the experimental group will receive 10 minutes before the procedure 1 g of tranexamic acid in 100 ml of saline intravenously unlike the patients in the control group who will receive just sterile saline.
  Arms: Tranexamic acid injectable product
Drug: Placebo — Patients from experimental group will receive 10 minutes before the procedure 1 g of tranexamic acid in 100 ml of saline intravenously unlike the patients in the control group who will receive just sterile saline.
  Arms: Placebo

SUMMARY:
Shoulder arthroscopy provides many benefits with a permanent increase in the possibilities and complexity of the application. A condition to perform it is intraoperative visual clarity dependent on hemorrhage control. The aim of this prospective, double blind, randomized, and controlled study is to examine the effect of intravenously administered tranexamic acid (TXA) on the visual clarity, perioperative hemorrhage, duration and early postoperative course of shoulder arthroscopy in beach chair position, which is not yet available in the literature. In the tested and control group, the investigators measure hemoglobin (Hb) in the waste irrigation fluid and the patient's blood before and after the procedure, visual clarity, duration of the procedure, postoperative shoulder swelling, pain level and analgesic drug consumption. The research uses scientific methods to determine if there is a reasonable basis for introducing TXA into routine clinical use.

DETAILED DESCRIPTION:
All surgical procedures will be performed at the University orthopaedic and trauma hospital Lovran, Croatia. Upon arrival at the hospital, the patient's body weight and height will be recorded. One day before the procedure, the patient will have blood taken from a vein and a complete blood count will be analyzed. Immediately before the procedure, patients will receive regional infiltrative (interscalene block) and general anesthesia with airway protection by endotracheal tube or laryngeal mask. Patients in the experimental group will receive 1 g of tranexamic acid in 100 ml of sterile saline IV 10 min before the start of the procedure, while patients in the control group will receive only sterile saline. The position of the patients will be beach chair with the head in the protective helmet and the arm in the front traction of 2-3 kg. All patients will be operated on by the same surgeon (NM) with the usual equipment: 4.5 mm 30° arthroscopic lens, arthroscopic pump basically set to 50 mmHg with the possibility of pulse increase of pressure by 20 mmHg for 2 min as needed, radiofrequency ablator and arthroscopic shaver system. Tendon reconstructions and shoulder stabilization will be performed in the usual way with suture anchors. During the procedure, the visual clarity on the endoscope screen (Visual analog scale VAS range: 0 worst visual clarity - 10 best visual clarity) will be evaluated by the surgeon every 15 minutes and the screen will be photographed at the same time. Screen photos will be presented after surgery to three independent surgeons with experience in arthroscopy on visual clarity estimation (VAS range 0-10). During the procedure, the number of times the pump pressure is increased will be counted. At the end of the surgery, the mean arterial pressure (MAP) will be noted, the exact amount of irrigation fluid consumed and the duration of the procedure from the first incision to the last skin suture will be calculated. A homogenized sample will be taken from the total volume of the waste solution in which the Hb concentration will be determined by a spectrophotometer using the Cripps method (University of Rijeka, Medical Faculty; spectrophotometer Varian Cary 100 Bio 190-900 nm, resolution ≤ 0.189 nm, wavelength accuracy of ± 0.02 nm to ± 0.04 nm). On the first day after the surgery, the shoulder circumference will be measured at 3 typical sites and the level of pain will be noted (VAS range 0 no pain -10 the strongest pain). On the second day, the shoulder circumference measurement and estimation of the level of pain will be repeated. Also blood will be taken from a vein and complete blood count will be repeated. During the postoperative period, the amount and type of analgesic drugs administered and the length of hospitalization will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* rotator cuff tear
* instability of the glenohumeral joint
* instability of the acromioclavicular joint

Exclusion Criteria:

* allergy to tranexamic acid
* deep vein thrombosis
* congenital thrombophilia
* coagulopathy
* thromboembolic events last 12 months
* stroke or acute coronary syndrome last 3 months
* renal failure
* cirrhosis of the liver
* glaucoma or retinal vascular disorder
* chronic treatment with anticoagulant therapy
* uncontrolled hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Visual clarity on endoscope screen during shoulder arthroscopy | At the very beginning of the shoulder arthroscopy
  The surgeon will evaluate visual clarity using Visual analog scale range from 0 (worst visual clarity) -10 (best visual clarity) every 15 minutes during shoulder arthroscopy and screen will be photographed at the same time
Visual clarity on endoscope screen during shoulder arthroscopy | After 15 minutes since the beginning of the surgery
  The surgeon will evaluate visual clarity using Visual analog scale range from 0 (worst visual clarity) -10 (best visual clarity) every 15 minutes during shoulder arthroscopy and screen will be photographed at the same time
Visual clarity on endoscope screen during shoulder arthroscopy | After 30 minutes since the beginning of the surgery
  The surgeon will evaluate visual clarity using Visual analog scale range from 0 (worst visual clarity) -10 (best visual clarity) every 15 minutes during shoulder arthroscopy and screen will be photographed at the same time
Visual clarity on endoscope screen during shoulder arthroscopy | After 45 minutes since the beginning of the surgery
  The surgeon will evaluate visual clarity using Visual analog scale range from 0 (worst visual clarity) -10 (best visual clarity) every 15 minutes during shoulder arthroscopy and screen will be photographed at the same time
Visual clarity on endoscope screen during shoulder arthroscopy | After 60 minutes since the beginning of the surgery
  The surgeon will evaluate visual clarity using Visual analog scale range from 0 (worst visual clarity) -10 (best visual clarity) every 15 minutes during shoulder arthroscopy and screen will be photographed at the same time
Visual clarity on endoscope screen during shoulder arthroscopy | After 75 minutes since the beginning of the surgery
  The surgeon will evaluate visual clarity using Visual analog scale range from 0 (worst visual clarity) -10 (best visual clarity) every 15 minutes during shoulder arthroscopy and screen will be photographed at the same time
Visual clarity on endoscope screen during shoulder arthroscopy | After 90 minutes since the beginning of the surgery
  The surgeon will evaluate visual clarity using Visual analog scale range from 0 (worst visual clarity) -10 (best visual clarity) every 15 minutes during shoulder arthroscopy and screen will be photographed at the same time
Visual clarity on endoscope screen during shoulder arthroscopy | After 105 minutes since the beginning of the surgery
  The surgeon will evaluate visual clarity using Visual analog scale range from 0 (worst visual clarity) -10 (best visual clarity) every 15 minutes during shoulder arthroscopy and screen will be photographed at the same time
Visual clarity on endoscope screen during shoulder arthroscopy | After 120 minutes since the beginning of the surgery
  The surgeon will evaluate visual clarity using Visual analog scale range from 0 (worst visual clarity) -10 (best visual clarity) every 15 minutes during shoulder arthroscopy and screen will be photographed at the same time
Visual clarity on endoscope screen during shoulder arthroscopy | After 135 minutes since the beginning of the surgery
  The surgeon will evaluate visual clarity using Visual analog scale range from 0 (worst visual clarity) -10 (best visual clarity) every 15 minutes during shoulder arthroscopy and screen will be photographed at the same time
Visual clarity on endoscope screen during shoulder arthroscopy | After 150 minutes since the beginning of the surgery
  The surgeon will evaluate visual clarity using Visual analog scale range from 0 (worst visual clarity) -10 (best visual clarity) every 15 minutes during shoulder arthroscopy and screen will be photographed at the same time
Visual clarity on endoscope screen during shoulder arthroscopy | Through study completion, an average of 1 year
  Screen photos taken every 15 minutes during shoulder arthroscopy will be presented after surgery to three independent surgeons with experience in arthroscopy on visual clarity estimation using Visual analog scale range from 0 (worst visual clarity) -10 (best visual clarity)
Perioperative blood loss | Right after the surgery
  The investigators will measure hemoglobin (Hb mg/100 mL) in the waste irrigation fluid collected during the surgery
Perioperative blood loss | 1 day before the surgery
  The investigators will measure hemoglobin (Hb g/L) in the patient's blood before and after the procedure
Perioperative blood loss | 2nd day after the surgery
  The investigators will measure hemoglobin (Hb g/L) in the patient's blood before and after the procedure
Early postoperative course of shoulder arthroscopy | One day before the surgery
  The investigators will measure postoperative shoulder swelling. Shoulder circumference will be measured in centimeters (cm) at 3 typical sites one day before the surgery and 1st and 2nd day after the surgery
Early postoperative course of shoulder arthroscopy | 1st day after the surgery
  The investigators will measure postoperative shoulder swelling. Shoulder circumference will be measured in centimeters (cm) at 3 typical sites one day before the surgery and 1st and 2nd day after the surgery
Early postoperative course of shoulder arthroscopy | 2nd day after the surgery
  The investigators will measure postoperative shoulder swelling. Shoulder circumference will be measured in centimeters (cm) at 3 typical sites one day before the surgery and 1st and 2nd day after the surgery
Early postoperative course of shoulder arthroscopy | 1st postoperative day
  The investigators will measure postoperative pain level with Visual analog scale range from 0 (no pain) - 10 (the strongest pain)
Early postoperative course of shoulder arthroscopy | 2nd postoperative day
  The investigators will measure postoperative pain level with Visual analog scale range from 0 (no pain) - 10 (the strongest pain)
Early postoperative course of shoulder arthroscopy | During hospitalization (up to 7 days)
  The investigators will measure analgesic drug consumption (mg of peroral or injectable product of paracetamol)
Early postoperative course of shoulder arthroscopy | During hospitalization (up to 7 days)
  The investigators will measure analgesic drug consumption (mg of peroral or injectable product of ketoprofen)
Early postoperative course of shoulder arthroscopy | During hospitalization (up to 7 days)
  The investigators will measure analgesic drug consumption (mg of injectable product of metamizole)
Early postoperative course of shoulder arthroscopy | During hospitalization (up to 7 days)
  The investigators will measure analgesic drug consumption (mg of injectable product of tramadol)

SECONDARY OUTCOMES:
Difference in blood loss between different indications for performing shoulder arthroscopy | Right after the surgery
  The investigators will measure hemoglobin (Hb mg/100 mL) in the waste irrigation fluid collected during the different types of shoulder arthroscopy
Difference in blood loss between different indications for performing shoulder arthroscopy | 1 day before the surgery
  The investigators will measure hemoglobin (Hb g/L) in the patient's blood before and after the different types of shoulder arthroscopy
Difference in blood loss between different indications for performing shoulder arthroscopy | 2nd day after the surgery
  The investigators will measure hemoglobin (Hb g/L) in the patient's blood before and after the different types of shoulder arthroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Nikola Matejcic, MD, Principal Investigator — University orthopaedic and trauma hospital Lovran, Croatia
Locations (1):
- University orthopaedic and trauma hospital, Lovran, Primorje-Gorski Kotar County, Croatia

IPD SHARING:
Plan to Share IPD: Yes
There will be a limit of access only to patients names
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After 1.9.2023 for 3 years
Access Criteria: Contact principal investigator

REFERENCES:
- [Background] Liu YF, Hong CK, Hsu KL, Kuan FC, Chen Y, Yeh ML, Su WR. Intravenous Administration of Tranexamic Acid Significantly Improved Clarity of the Visual Field in Arthroscopic Shoulder Surgery. A Prospective, Double-Blind, and Randomized Controlled Trial. Arthroscopy. 2020 Mar;36(3):640-647. doi: 10.1016/j.arthro.2019.10.020. Epub 2019 Dec 20. PMID 31870749
- [Background] Ersin M, Demirel M, Buget MI, Edipoglu IS, Atalar AC, Ersen A. The effect of intravenous tranexamic acid on visual clarity during arthroscopic rotator cuff repair: A randomized, double-blinded, placebo-controlled pilot study. Acta Orthop Traumatol Turc. 2020 Nov;54(6):572-576. doi: 10.5152/j.aott.2020.19164. PMID 33423986
- [Background] Cripps CM. Rapid method for the estimation of plasma haemoglobin levels. J Clin Pathol. 1968 Jan;21(1):110-2. doi: 10.1136/jcp.21.1.110. No abstract available. PMID 5697326
- [Background] Parker JD, Lim KS, Kieser DC, Woodfield TBF, Hooper GJ. Is tranexamic acid toxic to articular cartilage when administered topically? What is the safe dose? Bone Joint J. 2018 Mar 1;100-B(3):404-412. doi: 10.1302/0301-620X.100B3.BJJ-2017-1135.R1. PMID 29589496
- [Background] Gao HL, Zhang JC, He Y, Zhai WT, Xiao LB, Shi Q. [Clinical study on the control of intra-articular hemorrhage by tranexamic acid after shoulder arthroscopy]. Zhongguo Gu Shang. 2020 Mar 25;33(3):238-41. doi: 10.12200/j.issn.1003-0034.2020.03.010. Chinese. PMID 32233251
- [Background] Bayram E, Yildirim C, Erturk AK, Yilmaz M, Atlihan D. Comparison of the efficacy of irrigation with epinephrine or tranexamic acid on visual clarity during arthroscopic rotator cuff repair: A double-blind, randomized-controlled study. Jt Dis Relat Surg. 2021;32(1):115-121. doi: 10.5606/ehc.2021.78393. Epub 2021 Jan 6. PMID 33463426
- [Background] Hartland AW, Teoh KH, Rashid MS. Clinical Effectiveness of Intraoperative Tranexamic Acid Use in Shoulder Surgery: A Systematic Review and Meta-analysis. Am J Sports Med. 2021 Sep;49(11):3145-3154. doi: 10.1177/0363546520981679. Epub 2021 Jan 21. PMID 33475421
- [Background] Belk JW, McCarty EC, Houck DA, Dragoo JL, Savoie FH, Thon SG. Tranexamic Acid Use in Knee and Shoulder Arthroscopy Leads to Improved Outcomes and Fewer Hemarthrosis-Related Complications: A Systematic Review of Level I and II Studies. Arthroscopy. 2021 Apr;37(4):1323-1333. doi: 10.1016/j.arthro.2020.11.051. Epub 2020 Dec 2. PMID 33278534
- [Background] Rodriguez-Merchan EC. Tranexamic acid is effective in decreasing postoperative intraarticular bleeding in arthroscopic knee surgery. Blood Coagul Fibrinolysis. 2020 Apr;31(3):175-178. doi: 10.1097/MBC.0000000000000895. PMID 31990755
- [Background] Kirsch JM, Bedi A, Horner N, Wiater JM, Pauzenberger L, Koueiter DM, Miller BS, Bhandari M, Khan M. Tranexamic Acid in Shoulder Arthroplasty: A Systematic Review and Meta-Analysis. JBJS Rev. 2017 Sep;5(9):e3. doi: 10.2106/JBJS.RVW.17.00021. PMID 28902659
- [Background] Goldstein M, Feldmann C, Wulf H, Wiesmann T. Tranexamic Acid Prophylaxis in Hip and Knee Joint Replacement. Dtsch Arztebl Int. 2017 Dec 1;114(48):824-830. doi: 10.3238/arztebl.2017.0824. PMID 29249226
- [Background] Ng W, Jerath A, Wasowicz M. Tranexamic acid: a clinical review. Anaesthesiol Intensive Ther. 2015;47(4):339-50. doi: 10.5603/AIT.a2015.0011. Epub 2015 Mar 23. PMID 25797505
- [Background] van Montfoort DO, van Kampen PM, Huijsmans PE. Epinephrine Diluted Saline-Irrigation Fluid in Arthroscopic Shoulder Surgery: A Significant Improvement of Clarity of Visual Field and Shortening of Total Operation Time. A Randomized Controlled Trial. Arthroscopy. 2016 Mar;32(3):436-44. doi: 10.1016/j.arthro.2015.08.027. PMID 26524933
- [Background] Weber SC, Abrams JS, Nottage WM. Complications associated with arthroscopic shoulder surgery. Arthroscopy. 2002 Feb;18(2 Suppl 1):88-95. doi: 10.1053/jars.2002.31801. PMID 11828349
- [Background] Memon M, Kay J, Gholami A, Simunovic N, Ayeni OR. Fluid Extravasation in Shoulder Arthroscopic Surgery: A Systematic Review. Orthop J Sports Med. 2018 May 14;6(5):2325967118771616. doi: 10.1177/2325967118771616. eCollection 2018 May. PMID 29785406
- [Background] Rains DD, Rooke GA, Wahl CJ. Pathomechanisms and complications related to patient positioning and anesthesia during shoulder arthroscopy. Arthroscopy. 2011 Apr;27(4):532-41. doi: 10.1016/j.arthro.2010.09.008. Epub 2010 Dec 24. PMID 21186092
- [Background] Avery DM 3rd, Gibson BW, Carolan GF. Surgeon-rated visualization in shoulder arthroscopy: a randomized blinded controlled trial comparing irrigation fluid with and without epinephrine. Arthroscopy. 2015 Jan;31(1):12-8. doi: 10.1016/j.arthro.2014.08.010. Epub 2014 Nov 6. PMID 25442659
- [Background] Nho SJ, Freedman KB, Bansal SL, Romeo AA, Bach BR Jr, Bush-Joseph CA, Turner DA, Cole BJ. The effect of radiofrequency energy on nonweight-bearing areas of bone following shoulder and knee arthroscopy. Orthopedics. 2005 Apr;28(4):392-9. doi: 10.3928/0147-7447-20050401-16. PMID 15887586
- [Background] Tuijthof GJ, de Vaal MM, Sierevelt IN, Blankevoort L, van der List MP. Performance of arthroscopic irrigation systems assessed with automatic blood detection. Knee Surg Sports Traumatol Arthrosc. 2011 Nov;19(11):1948-54. doi: 10.1007/s00167-011-1495-z. Epub 2011 Apr 9. PMID 21479643
- [Background] Tuijthof GJ, Dusee L, Herder JL, van Dijk CN, Pistecky PV. Behavior of arthroscopic irrigation systems. Knee Surg Sports Traumatol Arthrosc. 2005 Apr;13(3):238-46. doi: 10.1007/s00167-004-0573-x. Epub 2005 Jan 4. PMID 15630604
- [Background] Burkhart SS, Danaceau SM, Athanasiou KA. Turbulence control as a factor in improving visualization during subacromial shoulder arthroscopy. Arthroscopy. 2001 Feb;17(2):209-12. doi: 10.1053/jars.2001.22298. PMID 11172254
- [Background] Ampat G, Bruguera J, Copeland SA. Aquaflo pump vs FMS 4 pump for shoulder arthroscopic surgery. Ann R Coll Surg Engl. 1997 Sep;79(5):341-4. PMID 9326125
- [Background] Morrison DS, Schaefer RK, Friedman RL. The relationship between subacromial space pressure, blood pressure, and visual clarity during arthroscopic subacromial decompression. Arthroscopy. 1995 Oct;11(5):557-60. doi: 10.1016/0749-8063(95)90131-0. PMID 8534296
- [Background] Jensen KH, Werther K, Stryger V, Schultz K, Falkenberg B. Arthroscopic shoulder surgery with epinephrine saline irrigation. Arthroscopy. 2001 Jul;17(6):578-81. doi: 10.1053/jars.2001.23590. PMID 11447543
- [Background] Smith JJ, Porth CM, Erickson M. Hemodynamic response to the upright posture. J Clin Pharmacol. 1994 May;34(5):375-86. doi: 10.1002/j.1552-4604.1994.tb04977.x. PMID 8089249
- [Background] Li X, Eichinger JK, Hartshorn T, Zhou H, Matzkin EG, Warner JP. A comparison of the lateral decubitus and beach-chair positions for shoulder surgery: advantages and complications. J Am Acad Orthop Surg. 2015 Jan;23(1):18-28. doi: 10.5435/JAAOS-23-01-18. PMID 25538127